CLINICAL TRIAL: NCT02616068
Title: A Phase III, Randomized, Double Blind, Non-inferiority, Comparative Study of the New Transdermal Patch Dosage Form Containing Loxoprofen Sodium (100 mg) and Loxonin® (60 mg Tablet) for the Treatment of Acute Traumatic Injuries
Brief Title: Comparative Study of Loxoprofen Sodium Transdermal Patch and Loxonin® Tablets for the Treatment of Acute Trauma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo Brasil Farmacêutica LTDA (Industry)
Collaborators: Quintiles, Inc. (Industry); Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS600-A-L301 - Loxonin Tape
Record Dates: First submitted 2015-11-24; First posted 2015-11-26 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Trauma; Pain
MeSH Terms: conditions — Wounds and Injuries; Pain | interventions — Transdermal Patch; loxoprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- transdermal patch & placebo (Experimental): transdermal patch 100 mg once a day for 7 days and placebo (for loxoprofen sodium 60 mg tablet) by mouth, every 8 hours for 7 days
  Interventions: Drug: Transdermal Patch; Drug: Placebo (for loxoprofen sodium)
- loxoprofen sodium & placebo (Active Comparator): loxoprofen sodium 60 mg by mouth, every 8 hours for 7 days and placebo (for transdermal patch 100 mg) once a day for 7 days
  Interventions: Drug: Loxoprofen sodium; Drug: Placebo (for transdermal patch)

INTERVENTIONS:
Drug: Transdermal Patch — Transdermal patch 100 mg once a day for 7 days
  Arms: transdermal patch & placebo
Drug: Loxoprofen sodium — Loxoprofen sodium 60 mg per tablet by mouth, every 8 hours for 7 days
  Arms: loxoprofen sodium & placebo
Drug: Placebo (for loxoprofen sodium) — Placebo (for loxoprofen sodium 60 mg per tablet) by mouth, every 8 hours for 7 days
  Arms: transdermal patch & placebo
Drug: Placebo (for transdermal patch) — Placebo (for transdermal patch 100 mg) once a day for 7 days
  Arms: loxoprofen sodium & placebo

SUMMARY:
This study evaluates the non-inferiority of the new transdermal patch dosage form containing loxoprofen sodium (100 mg - Daiichi-Sankyo) in comparison with oral Loxonin® (60 mg tablet - Daiichi-Sankyo) for the treatment of acute traumatic injuries.

DETAILED DESCRIPTION:
The primary objective of the study will be to verify the efficacy of loxoprofen in its new dosage form for the treatment of pain.

Primary endpoint: score of change in spontaneous pain by using the visual analogue scale (VAS) after seven days of treatment.

Secondary endpoints: intensity of pain evaluated by the VAS scale on each study visit, impression of the research subject checked by a 7-point scale, changes in clinical symptoms, and frequency of use of the rescue medication. Evaluation of drug safety as per the occurrence of adverse events and serious adverse events.

This is a double blind, randomized, comparative study, with a total of 208 subjects divided into 2 groups: 104 subjects treated with loxoprofen sodium (transdermal patch 100 mg; Daiichi-Sankyo) associated with placebo tablet (experimental group) and 104 subjects treated with transdermal patch of placebo associated with Loxonin® (loxoprofen sodium 60 mg - Daiichi-Sankyo - control group).

In order to be enrolled in the study, the research subject shall sign and date the informed consent form and shall have between 18 and 65 years old, with recent (48 hours before study baseline visit) posttraumatic disease (contusion or sprain) of lower or upper limbs (except for fingers and toes), with at least one moderate or more serious symptom of pain or inflammation according to the investigator's evaluation, with no prior (5 days before initiating the study treatment) or current use of pain medication, NSAIDs, anti-inflammatory drugs, or steroids. In addition, research subjects shall not experience cardiovascular, renal, or hematological diseases, diabetes mellitus, psychiatric disorders, or any other serious comorbidity (at the investigator's discretion), apparent complication of a bacterial infection, fracture or requiring immobilization with cast or surgical procedure, neck sprain, too small area affected (e.g.,fingers) not allowing the use of the transdermal patch, skin sores in application site, bad or sensitive condition of the skin with prior history of dermatitis due to the use of topic drugs, prior history of gastrointestinal bleeding or ulcers, bronchial asthma of any cause, allergy to loxoprofen or any other NSAIDs. Also, the subjects should not have participated in any other clinical study in the last 12 months and pregnant or breastfeeding subjects or those who want to become pregnant or who refuse to use a safe birth control method during the study will not be enrolled in the study.

The accrual period anticipated for the study will be of 4 to 5 months as of the regulatory approval of the protocol. Total duration of participation of each research subject and active treatment will be of 1 week.

ELIGIBILITY:
Inclusion Criteria:

* For enrollment in this study, the eligible research subjects shall meet all criteria below:

  * Sign and date the informed consent form;
  * Age between 18 and 65 years old;
  * Have recent (48 hours before study baseline visit) post-traumatic disease (contusion or sprain) of lower or upper limbs (except for fingers and toes), with at least one moderate or more serious symptom of pain or inflammation according to the investigator's evaluation.

Exclusion Criteria:

* Research subjects who meet any criteria below will not be eligible for the study:

  * Have cardiovascular, renal, or hematological disease, diabetes mellitus, gastrointestinal disease, hepatic disease, asthma, rheumatoid arthritis, osteoarthritis, or any other serious chronic comorbidity (at the investigator's discretion);
  * Prior history of gastrointestinal bleeding or ulcers (6 months before enrollment in the study);
  * Have any hemorrhagic disorder;
  * Have apparent complication of bacterial infection;
  * Have a fracture or need of immobilization with cast or surgical procedure or neck sprain;
  * Have a too small area affected (e.g., fingers) not allowing the use of the transdermal patch, skin sores in application site, bad or sensitive condition of the skin with prior history of dermatitis due to the use of topic drugs;
  * Have made a prior (5 days before the study treatment is initiated) or current use of pain medications, NSAIDs, anti-inflammatory drugs, or steroids;
  * Have a known allergy to loxoprofen, inactive ingredients of the formulation or any other NSAIDs;
  * Subjects who are pregnant or breastfeeding or those who want to become pregnant or who refuse to use a safe birth control method during the study;
  * Research subjects who have participated in another clinical study in the last 12 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Score of change in spontaneous pain by using the visual analogue scale (VAS) | after seven days of treatment.

SECONDARY OUTCOMES:
Intensity of pain evaluated by the VAS scale | on day 3 and on day 7
Impression of the research subject checked by a 7-point scale | on day 3 and on day 7
Evaluation of drug safety as per the occurrence of adverse events and serious adverse events. | on day 3 and on day 7, for SAE up to 30 days

CONTACTS AND LOCATIONS:
Locations (8):
- Brazil (8):
  - Ctd Clinica de Terapia Da Dor Ltda, Salvador, Estado de Bahia
  - Med Centro de Estudos- Crd- Centro, Goiânia, Goiás
  - CMiP - Centro Mineiro de Pesquisa, Juiz de Fora, Minas Gerais
  - Hospital São Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - HMCG - Hospital e Maternidade Dr. Christovão da Gama, Santo André, São Paulo
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - Hospital Nipo-Brasileiro, São Paulo, São Paulo

REFERENCES:
- [Background] Dreiser RL. Topical antirheumatic drug therapy: current practice and future trends. Eur J Rheumatol Inflamm. 1994;14(4):3-8. No abstract available. PMID 7601180
- [Result] Garrett WE Jr. Muscle strain injuries: clinical and basic aspects. Med Sci Sports Exerc. 1990 Aug;22(4):436-43. PMID 2205779
- [Result] Liu SH, Nguyen TM. Ankle sprains and other soft tissue injuries. Curr Opin Rheumatol. 1999 Mar;11(2):132-7. doi: 10.1097/00002281-199903000-00009. PMID 10319217
- [Result] Almekinders LC. Anti-inflammatory treatment of muscular injuries in sport. An update of recent studies. Sports Med. 1999 Dec;28(6):383-8. doi: 10.2165/00007256-199928060-00001. PMID 10623981
- [Result] Jarvinen TA, Jarvinen TL, Kaariainen M, Kalimo H, Jarvinen M. Muscle injuries: biology and treatment. Am J Sports Med. 2005 May;33(5):745-64. doi: 10.1177/0363546505274714. PMID 15851777
- [Result] Garrett WE Jr, Nikolaou PK, Ribbeck BM, Glisson RR, Seaber AV. The effect of muscle architecture on the biomechanical failure properties of skeletal muscle under passive extension. Am J Sports Med. 1988 Jan-Feb;16(1):7-12. doi: 10.1177/036354658801600102. PMID 3344884
- [Result] Garrett WE Jr, Safran MR, Seaber AV, Glisson RR, Ribbeck BM. Biomechanical comparison of stimulated and nonstimulated skeletal muscle pulled to failure. Am J Sports Med. 1987 Sep-Oct;15(5):448-54. doi: 10.1177/036354658701500504. PMID 3674268
- [Result] Arrington ED, Miller MD. Skeletal muscle injuries. Orthop Clin North Am. 1995 Jul;26(3):411-22. PMID 7609956
- [Result] Classification of chronic pain. Descriptions of chronic pain syndromes and definitions of pain terms. Prepared by the International Association for the Study of Pain, Subcommittee on Taxonomy. Pain Suppl. 1986;3:S1-226. No abstract available. PMID 3461421
- [Result] Carr DB, Goudas LC. Acute pain. Lancet. 1999 Jun 12;353(9169):2051-8. doi: 10.1016/S0140-6736(99)03313-9. PMID 10376632
- [Result] Stanos SP. Topical agents for the management of musculoskeletal pain. J Pain Symptom Manage. 2007 Mar;33(3):342-55. doi: 10.1016/j.jpainsymman.2006.11.005. PMID 17349504